CLINICAL TRIAL: NCT04103255
Title: High Frequency Multimodal Training Including Tai Chi for Improving Motor and Cognitive Function in People With Parkinson's Disease
Brief Title: High Frequency and Intensive Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Parkinson Schweiz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BSL prevention program
Record Dates: First submitted 2019-09-17; First posted 2019-09-25 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
Keywords: Cognition; Tai Chi
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency and intensive prevention (Experimental): High frequency and intensive prevention program
  1. Tai Chi
  2. CogniFit (cognitive training)
  3. SpeechCare (speech training)
  Interventions: Other: High frequency and intensive prevention program
- Control group (CogniPlus) (Active Comparator): Computer-assisted cognitive training program
  Interventions: Other: High frequency and intensive prevention program

INTERVENTIONS:
Other: High frequency and intensive prevention program — This study is a 4 week non-randomized controlled trial (RCT)

SUMMARY:
The treatment of PD has made considerable advances in recent years with respect to drug therapies, as well as many new physiotherapy and drug-based methods, and there have also been great improvements in therapy thanks to deep brain stimulation. Cognitive rehabilitation has shown to be effective in PD (Abbruzzese et al., 2016), however, there has yet to be a major breakthrough in the treatment and prevention of PDD (Parkinson's Disease Dementia ). This is where the high frequency and intensive prevention described here comes into play.

DETAILED DESCRIPTION:
Cognitive decline is an important and common complication in Parkinson's Disease (PD); approximately 27% of non-demented PD patients have Mild Cognitive Impairment (MCI) (Litvan et al. 2012, Chaudhuri et al., 2011) and up to 80% develop PD dementia (PD-D) over the long term (Hely et al., 2005). Cognitive course in PD is heterogeneous and affects visuospatial, attentional, executive and memory function; studies report different cognitive subtypes and divergent patterns of cognitive decline (Kehagia et al., 2010; Litvan et al., 2011; Williams-Gray et al., 2007; Yarnall et al., 2014). Recently, models have been constructed to estimate individual risk for global cognitive impairment using a small set of predictor variables (Liu et al. 2017; Velseboer et al., 2016). These prediction algorithms were developed in large samples of PD patients and accurately forecast cognitive decline in both, patients with MCI and patients with PD-D and were successfully replicated in independent samples; a score with a predefined cut off point predicts dementia with high positive and negative predictive values (Liu et al., 2017).

The primary aim of this study is the possible stabilization or delay of cognitive decline as well as the improvement of the quality of life of the patients. As secondary outcome, the change in symptoms associated with PD, will be investigated. Psychological states as depression and anxiety, as well as cognitive performance in different areas, for example attention and memory shall be investigated. Neurological symptoms, for example motor function and sleepiness, will also be assessed as secondary parameters and potentially confounding factors.

This study is a 4 week non-randomized controlled trial with one intervention group (HIPP) and one control group (CogniPlus). Primary and secondary outcome measures are assessed at baseline and are repeated after the 4-week intervention period and at 6 month in a follow-up assessment. After 4 weeks there is an intermediate measurement consisting of the primary outcome measures.

The intervention group receives individualized program: the program will be tailored to the patient's needs, strengths and weaknesses, resulting from the initial assessment.

1. Tai Chi - "Keep Moving" is an exercise programme for patients with movement disorders that explicitly utilizes the health aspect of Tai Chi movement teachings. Each session lasted 60 minutes and ended with a 10-minute meditation. The Tai Chi sessions in our study were carried out twice a week under the guidance of certified Tai Chi instructors. Details of this program can be found on the following website: https://taiji-therapie.ch/
2. CogniFit® - is a online-based personalized cognition training program. This well-validated cognitive training improves attention, working memory, memory, executive function, and visual perceptual functions. Each session lasted 20 minutes and was applied 2-5 times per week based on the results of the baseline tests. The home-based approach took place under the supervision of a psychologist or a specially trained psychology student. The difficulty level was automatically adjusted by the program itself. Details of the program can be found on the following website: https://www.cognifit.com/.
3. SpeechCare - (MoveApp) is a home-based approach for patients with Parkinson's disease. The training program uses automatic speech recognition (ASR) and thus can provide feedback on speech intelligibility. Each session lasted 12 minutes and was conducted 1-3 times per week based on the results of the baseline test of SpeechCare . The domestic approach took place under the supervision of a psychologist or a specially trained psychology student. The level of difficulty was manually adjusted as needed. Details of the program can be found on the following website: https://www.speechcare.de/.

The patients in the control group received a computer-assisted cognitive training program: CogniPlus (Schuhfried GmbH, Vienna, Austria). Each training session consisted of different tasks (Focused attention; working memory; planning and action skill; respons inhibition) that were performed for 10 Minutes each. Details of the program can be found on the following website: www.schuhfried.at. The training sessions were supervised by a psychologist or a specially trained student of psychology

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson syndrome according to United Kingdom Parkinson's Disease Brain Bank Criteria
* mental competence to provide informed consent
* able to understand German sufficiently

Exclusion Criteria:

* Severe dementia (DMS-IV, mini mental Status (MMS) <24, moca test (MoCa) <21)
* young onset Parkinson's disease (<18y)
* other neurological or psychiatric diseases of the brain not related to PD
* secondary parkinsonism
* physical impairment hindering the adequate execution of the training
* insufficient knowledge of German
* pregnancy
* Deep Brain Stimulation (DBS) is no exclusion criterion.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Episodic memory: California Verbal Learning Test (CVLT; Delis, Kramer, Ober, & Kaplan, 1987) | Before and after 4 weeks of training, After 6-month
  This is a method that tests memory functions, including encoding, retrieval, and recognition processes. The task is to learn in five cycles a shopping list of 16 words assigned to four semantic categories (i.e. beverages, fruits, clothing, tools). As many words as possible should be enumerated after each cycle. The sum of the words stored in the 1-5 cycles is used as the encoding parameter.
working memory: Corsi Block Test (Härtig et al., 2000) | Before and after 4 weeks of training, After 6-month
  Corsi Block Test serve to evaluate the verbal and visual working memory. In the Corsi Block, the test person is presented with a board with irregularly arranged cubes. The task is to remember a sequence of tapped cubes and then to tap the cubes in the same sequence or later to follow the path shown in reverse order. Also with this test the difficulty increases, as the offered sequences become increasingly longer.
  The total score for the Digit Span is the sum of 12 items, ranging from 0 (worst possible result) to 12 (best possible result).
  The total score for the Corsi Block is the sum of 14 points in forward typing, ranging from 0 (worst score) to 14 (best symptoms) and the sum of 12 points in backward typing from 0 (worst score) to 12 (best symptoms).
Visuo-construction: Rey-Osterrieth complex figure (Duley et al., 1993) | Before and after 4 weeks of training, After 6-month
  The Rey-Osterrieth (ROCF) and Taylor (TCF) complex figure tests are widely used to assess visuospatial and constructional abilities as well as visual/non-verbal Memory (Marie-Pier Tremblay et al., 2015). The score ranging from 0 (worst possible result) to 36 (best possible result).
  ·
Attention: Trail Making Test, part A (J. Perianez et al., 2007) | Before and after 4 weeks of training, After 6-month
  Trail Making Test, part A serve to evaluate the attention
Executive function (flexibility): Wisconsin Card Sorting test, number of errors (H.E. Nelson, 1976) | Before and after 4 weeks of training, After 6-month
  Wisconsin Card Sorting test serve to evaluate the executive function

SECONDARY OUTCOMES:
Electroencephalogram (EEG) | Before and after 4 weeks of training, After 6-month
  1. EEG power in Delta; Theta; Alpha 1; Alpha 2; Beta.
  2. Brain Network Connectivity
Near-infrared spectroscopy | Before and after 4 weeks of training, After 6-month
  Detecting changes in blood hemoglobin concentrations associated with neural activity
Unified Parkinson's Disease Rating Scale UPDRS Part III | Before and after 4 weeks of training, After 6-month
  This is the standard scale used for grading severity of PD. (UPDRS) - Four Parts Higher score values represent a worse outcome.
  Part I: Mentation, Behavior and Mood - 4 questions 1-4 Score range: 1-16; Part II: Activities of Daily Living - 13 questions 5-17 Score range: 0-52 Part III: Motor Examination - 19 questions 18-31 and 25 total assessments Score range: 0-100 Part IV: Complications of Therapy (In the past week) - 11 questions Score range: 0-25
Tinetti Mobility Test (D.A. Kegelmeyer et al., 2007) | Before and after 4 weeks of training, After 6-month
  Balance and stability assessment
Epworth Sleepiness Scale (M.W. Johns, 1991) | Before and after 4 weeks of training, After 6-month
  Measuring Daytime Sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, Prof.Dr.med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Toloraia K, Gschwandtner U, Fuhr P. High-frequency multimodal training with a focus on Tai Chi in people with Parkinson's disease: a pilot study. Front Aging Neurosci. 2024 Feb 15;16:1335951. doi: 10.3389/fnagi.2024.1335951. eCollection 2024. PMID 38425785